CLINICAL TRIAL: NCT03851991
Title: A 52-week Multicenter, Randomized, Double-blind, Placebo-controlled, Prospective Study to Evaluate the Efficacy and Safety of Arbidol in Reducing the Frequency of AECOPD.
Brief Title: The Efficacy and Safety of Arbidol in Reducing the Frequency of AECOPD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, LI ZHAO, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX002
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: COPD Patients
Keywords: AECOPD; Arbidol
MeSH Terms: interventions — umifenovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arbidol (Active Comparator): 200mg, three times per day, for 2-5 Days.
  Interventions: Drug: Arbidol
- control (Placebo Comparator): two capsules, three times per day, for 2-5 Days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Arbidol — oral
  Arms: arbidol
Drug: Placebos — controle
  Arms: control

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is currently the fourth leading cause of death in the world. Acute exacerbations of COPD (AECOPD) are the most important events in the course of the disease because they negatively impact health status, life quality, disease progression, patients survival and economic and social burden. Reducing frequency of AECOPD is the key goal of management for COPD. Since respiratory viral infections are the mainly trigger of AECOPD, anti-viral therapy would be the affective method to prevent the exacerbation or reduce the attack severity. However, there are no positive study results of treating or preventing AECOPD used by current anti-viral drugs approved by FDA so far.

Arbidol is a non-nucleoside antiviral drug. It inhibits viral DNA and RNA synthesis by inhibiting fusion of viral lipid vesicle membrane with host cell membranes. Arbidol has broad-spectrum antiviral activity. In addition to inhibition of influenza virus, it against a variety of viruses including respiratory syncytial disease (RSV), parainfluenza virus, human rhinovirus, coxsackie virus (CV), adenovirus (ADV) and so on. In recent years, some fundamental and clinical researches have shown that arbidol has a significant role in prevention and treatment of influenza virus and other acute respiratory viral infections. Therefore, the investigators speculate that Arbidol will effectively control COPD combined with upper respiratory virus infection, thereby reducing acute exacerbations of COPD.

This is a prospective, multicenter, randomized, double-blind, placebo-controlled, 52-week study. The purpose of this study is to evaluate the efficacy and safety of arbidol in improving the frequency and extent of moderate or severe acute exacerbations in patients with COPD. Eligible subjects will be randomly assigned to treatment group or placebo group at a 2:1 ratio. Subjects of treatment group receive an on-demand arbidol 200 mg three times per day while placebo group receives matched placebo. When the subject has a new respiratory infection, original respiratory symptoms worsen, or fever (the lower body temperature is greater than 37.3℃), oral medication is given immediately. The subjects are required to receive the first dose of drug within 8 hours after the symptoms of upper respiratory tract infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from Outpatient clinic.
2. Informed consent and assent must be obtained before any study assessment is performed.
3. Aged ≥40 years.
4. Continuous respiratory symptoms, such as chronic cough, sputum or shortness of breath etc.
5. Exposure to risk factors: Host factors, Tobacco, Occupation, Indoor/outdoor pollution
6. FEV1/FVC less than 0.70 after withholding bronchodilator.
7. 2 or more acute exacerbations of COPD within the 12 months prior to visit 0. Or more than 1 hospitalizations due to AECOPD within the 12 months prior to visit 0.
8. Good compliance.

Exclusion Criteria:

1. Patients with any chronic diseases except COPD which in the opinion of the investigator may interfere with study evaluation or optimal participation in the study.
2. Patients with a history of chronic lung disease other than COPD, including (but not limited to) active tuberculosis, lung cancer, clinically significant bronchiectasis, primary pulmonary hypertension, sarcoidosis, interstitial lung disease, asthma (other than asthma COPD overlap), severe cor pulmonale.
3. Patients with acute coronary syndrome(ACS) or acute left heart failure within the 6 months prior to visit 0. Patients accepted Coronary interventional therapy or coronary artery bypass grafting due to ACS within the 3 months prior to visit 0.
4. Patients with uncontrolled hypertension.
5. Patients who started oral >10mg prednisolone or Equivalent systemic corticosteroids within 4 weeks prior to Visit 1. Or patients who received antibiotics within 4 weeks prior to Visit 1. Or patients who received standard treatment for COPD within 4 weeks prior to Visit 1. Or use of other investigational drugs within 5 half-lives of enrollment, or within 30 days, whichever is longer.
6. Patients who received influenza vaccine or other viral vaccine within the 12 months prior to visit 0.
7. The end of AECOPD therapy was within the 4 weeks prior to visit 0. Or Occurrence of AECOPD within the 6 weeks prior to visit 0.
8. History of arbidol sensitivity.
9. No person directly associated with the administration of the study is allowed to participate as a study subject.
10. Use of other investigational intervention within within 30 days.
11. Patients with obviously abnormal liver function, AST or ALT>2 times the upper limit of normal value or total bilirubin>1.3 times the upper limit of normal value.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Frequency of moderate or severe acute exacerbation in patients with chronic obstructive pulmonary disease | 52 weeks
  Frequency of moderate or severe acute exacerbation in patients with chronic obstructive pulmonary disease

SECONDARY OUTCOMES:
The frequency of Acute exacerbation of patients leads to hospitalization | 52 weeks
  The frequency of Acute exacerbation of patients leads to hospitalization
The intervals to the next acute exacerbation after the first use of the study drug | 52 weeks
  The intervals to the next acute exacerbation after the first use of the study drug
To assess the change of FEV1 from baseline | 52 weeks
  To assess the change of FEV1 from baseline
Mean duration of moderate or severe acute exacerbation in chronic obstructive pulmonary disease | 52 weeks
  Mean duration of moderate or severe acute exacerbation in chronic obstructive
Throat swab and virus separation experiment to detect the composition of respiratory viruses in patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) requiring hospitalization | 52 weeks
  Throat swab and virus separation experiment to detect the composition of respiratory viruses in patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) requiring hospitalization
Number of unscheduled visits to a clinic for COPD exacerbation | 52 weeks
  Number of unscheduled visits to a clinic for COPD exacerbation
Number of emergency room visits for AECOPD | 52 weeks
  Number of emergency room visits for AECOPD
Number of hospitalizations due to AECOPD | 52 weeks
  Number of hospitalizations due to AECOPD

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhao, Doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko FW, Chan KP, Hui DS, Goddard JR, Shaw JG, Reid DW, Yang IA. Acute exacerbation of COPD. Respirology. 2016 Oct;21(7):1152-65. doi: 10.1111/resp.12780. Epub 2016 Mar 30. PMID 27028990
- [Background] Zwaans WA, Mallia P, van Winden ME, Rohde GG. The relevance of respiratory viral infections in the exacerbations of chronic obstructive pulmonary disease-a systematic review. J Clin Virol. 2014 Oct;61(2):181-8. doi: 10.1016/j.jcv.2014.06.025. Epub 2014 Jul 4. PMID 25066886
- [Background] Brooks MJ, Burtseva EI, Ellery PJ, Marsh GA, Lew AM, Slepushkin AN, Crowe SM, Tannock GA. Antiviral activity of arbidol, a broad-spectrum drug for use against respiratory viruses, varies according to test conditions. J Med Virol. 2012 Jan;84(1):170-81. doi: 10.1002/jmv.22234. Epub 2011 Oct 25. PMID 22028179